CLINICAL TRIAL: NCT03961646
Title: Evaluation of the FOCUS Diffusion's Added Clinical Value Compared to Conventional MRI With Wide Field View Diffusion in Focal Pancreatic Lesions Characterization
Brief Title: Evaluation of the FOCUS Diffusion's Added Clinical Value Compared to Conventional MRI
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: Diffusion Focus
Record Dates: First submitted 2019-05-22; First posted 2019-05-23 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Cancer of Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The radiologist plays a key role in the management of pancreatic tumours, which are potentially serious.

While the scanner, with its high spatial resolution, plays a major role in pancreatic pathology, and in particular in the assessment of operability, MRI, with its good contrast resolution, has proven its contribution to the detection and characterization of focal lesions.

Each MRI examination consists of several series of images called sequences, each with its own particularity, to highlight different types of abnormalities such as edema, bleeding, tumor content or vascularization. All the sequences performed constitute a "protocol". The diffusion sequence is a technology that allows the microscopic random movements of water molecules to be translated into images. It thus makes it possible to differentiate between certain aggressive tumours which are characterised by a higher cell density than healthy tissue, in which water molecules do not circulate freely, benign lesions such as cysts in which the circulation of water molecules is not hindered. The calculation of the Apparent Diffusion Coefficient (ADC), an estimate of the diffusion rate of water molecules, is a quantitative diagnostic tool validated in many fields of application and in particular in oncology.

DETAILED DESCRIPTION:
This diffusion sequence has shown its usefulness in pancreatic pathology in the detection and characterization of focal pancreatic lesions, particularly for neuroendocrine tumors, the evaluation of chronic and autoimmune pancreatitis or the early detection of malignant transformation of certain high-risk cystic lesions. The diffusion sequence usually performed is called "wide field" because it covers the entire abdomen. The radiologist can thus analyse the neighbouring organs and in particular the liver, which makes it essential when a pancreatic tumour is suspected because of the risk of liver metastases.

This wide-field sequence suffers from several limitations: difficulty in differentiating adenocarcinomas from chronic pseudo-mass pancreatitis due to the overlap of CDA values and difficulty in defining the boundaries of cephalic or corporal adenocarcinomas due to the hypersignal of upstream chronic obstructive pancreatitis (9)(10). Technically, it is subject to movement artifacts related to respiration, adjacent organs and in particular the duodenum, and to an average spatial resolution of the pancreas.

Over the last 10 years, a diffusion sequence called "FOCUS" has been developed allowing a reduction of the field of view in the direction of phase coding and therefore a "zoomed" image with higher resolution. This sequence has shown interest in neuroradiology and prostate cancer detection in reducing artifacts and achieving better spatial resolution than the usual "wide field" diffusion sequence. 3 minutes and 30 seconds more are required to complete this sequence.

The pancreas is a good candidate for FOCUS diffusion imaging because of its small size, susceptibility to movement artifacts and spatial orientation, allowing antero-posterior reduction of the field of view. Initial work has established the feasibility of this FOCUS diffusion in pancreatic imaging and shown an improvement in image quality (more accurate and less artefacts) in FOCUS diffusion compared to the usual "wide field".

Due to its potential in pancreatic imaging, the FOCUS diffusion sequence has been performed in current practice since 2014 in the imaging department of the Groupe Hospitalier Paris Saint-Joseph (GHPSJ) in addition to the "wide field" diffusion sequence. The protocol thus created is called "combined protocol" as opposed to "standard protocol" which does not contain the FOCUS broadcast sequence.

Kim H et al showed an improvement in the subjective clinical utility of readers in the diagnosis of benign or malignant pancreatic lesions. However, it should be noted that in this study the authors compared the two sequences by opposing them rather than comparing the usual wide-field sequence with the combination of the two sequences.

ELIGIBILITY:
Inclusion Criteria:

* Male or female whose age ≥ 18 years old (Adult patient)
* Francophone patient
* Pancreatic MRI performed at the GHPSJ on 3 Tesla MRI between September 2014 (date of introduction of the FOCUS diffusion sequence) and April 2018
* Presence of at least one proven benign or malignant focal pancreatic lesion visible on at least one of the MRI sequences

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient objecting to the use of their data for this research
* Papillary and mucinous intra-channel tumour of pancreas (TIPMP) of secondary channels measuring less than 30mm.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with benign or malignant pancreatic lesions.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | Time of inclusion
  Diagnostic accuracy difference between the standard protocol and the combined protocol.

SECONDARY OUTCOMES:
Diagnostic performances of benignity or malignancy | Time of inclusion
  Differences between the standard protocol and the combined protocol in terms of sensitivity and specificity in the diagnosis of benign or malignant tumors.
Diagnostic confidence of radiologist's benign or malignant condition | Time of inclusion
  Confidence scores assigned by radiologist
Lesions' detected number | Time of inclusion
  Differences between the FOCUS diffusion sequence and the "wide field" sequence in terms of lesions' detected number
Image quality | Time of inclusion
  Differences between the FOCUS diffusion sequence and the "wide field" sequence in terms of image quality

CONTACTS AND LOCATIONS:
Overall Officials: Marc ZINS, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Schima W. MRI of the pancreas: tumours and tumour-simulating processes. Cancer Imaging. 2006 Dec 20;6(1):199-203. doi: 10.1102/1470-7330.2006.0035. PMID 17208676
- [Background] Koh DM, Collins DJ. Diffusion-weighted MRI in the body: applications and challenges in oncology. AJR Am J Roentgenol. 2007 Jun;188(6):1622-35. doi: 10.2214/AJR.06.1403. PMID 17515386
- [Background] Barral M, Taouli B, Guiu B, Koh DM, Luciani A, Manfredi R, Vilgrain V, Hoeffel C, Kanematsu M, Soyer P. Diffusion-weighted MR imaging of the pancreas: current status and recommendations. Radiology. 2015 Jan;274(1):45-63. doi: 10.1148/radiol.14130778. PMID 25531479
- [Background] Park MJ, Kim YK, Choi SY, Rhim H, Lee WJ, Choi D. Preoperative detection of small pancreatic carcinoma: value of adding diffusion-weighted imaging to conventional MR imaging for improving confidence level. Radiology. 2014 Nov;273(2):433-43. doi: 10.1148/radiol.14132563. Epub 2014 Jul 4. PMID 24991989
- [Background] d'Assignies G, Fina P, Bruno O, Vullierme MP, Tubach F, Paradis V, Sauvanet A, Ruszniewski P, Vilgrain V. High sensitivity of diffusion-weighted MR imaging for the detection of liver metastases from neuroendocrine tumors: comparison with T2-weighted and dynamic gadolinium-enhanced MR imaging. Radiology. 2013 Aug;268(2):390-9. doi: 10.1148/radiol.13121628. Epub 2013 Mar 26. PMID 23533288
- [Background] Motosugi U, Ichikawa T, Morisaka H, Sou H, Muhi A, Kimura K, Sano K, Araki T. Detection of pancreatic carcinoma and liver metastases with gadoxetic acid-enhanced MR imaging: comparison with contrast-enhanced multi-detector row CT. Radiology. 2011 Aug;260(2):446-53. doi: 10.1148/radiol.11103548. Epub 2011 Jun 21. PMID 21693662
- [Background] Kim HW, Lee JC, Paik KH, Kang J, Kim YH, Yoon YS, Han HS, Kim J, Hwang JH. Adjunctive role of preoperative liver magnetic resonance imaging for potentially resectable pancreatic cancer. Surgery. 2017 Jun;161(6):1579-1587. doi: 10.1016/j.surg.2016.12.038. Epub 2017 Feb 23. PMID 28237643
- [Background] Zins M, Matos C, Cassinotto C. Pancreatic Adenocarcinoma Staging in the Era of Preoperative Chemotherapy and Radiation Therapy. Radiology. 2018 May;287(2):374-390. doi: 10.1148/radiol.2018171670. PMID 29668413
- [Background] Klauss M, Lemke A, Grunberg K, Simon D, Re TJ, Wente MN, Laun FB, Kauczor HU, Delorme S, Grenacher L, Stieltjes B. Intravoxel incoherent motion MRI for the differentiation between mass forming chronic pancreatitis and pancreatic carcinoma. Invest Radiol. 2011 Jan;46(1):57-63. doi: 10.1097/RLI.0b013e3181fb3bf2. PMID 21139505
- [Background] Wiggermann P, Grutzmann R, Weissenbock A, Kamusella P, Dittert DD, Stroszczynski C. Apparent diffusion coefficient measurements of the pancreas, pancreas carcinoma, and mass-forming focal pancreatitis. Acta Radiol. 2012 Mar 1;53(2):135-9. doi: 10.1258/ar.2011.100252. Epub 2012 Jan 19. PMID 22262868
- [Background] Bittencourt LK, Matos C, Coutinho AC Jr. Diffusion-weighted magnetic resonance imaging in the upper abdomen: technical issues and clinical applications. Magn Reson Imaging Clin N Am. 2011 Feb;19(1):111-31. doi: 10.1016/j.mric.2010.09.002. PMID 21129638
- [Background] Saritas EU, Cunningham CH, Lee JH, Han ET, Nishimura DG. DWI of the spinal cord with reduced FOV single-shot EPI. Magn Reson Med. 2008 Aug;60(2):468-73. doi: 10.1002/mrm.21640. PMID 18666126
- [Background] Andre JB, Zaharchuk G, Saritas E, Komakula S, Shankaranarayan A, Banerjee S, Rosenberg J, Nishimura DG, Fischbein NJ. Clinical evaluation of reduced field-of-view diffusion-weighted imaging of the cervical and thoracic spine and spinal cord. AJNR Am J Neuroradiol. 2012 Nov;33(10):1860-6. doi: 10.3174/ajnr.A3134. Epub 2012 May 3. PMID 22555576
- [Background] Reischauer C, Wilm BJ, Froehlich JM, Gutzeit A, Prikler L, Gablinger R, Boesiger P, Wentz KU. High-resolution diffusion tensor imaging of prostate cancer using a reduced FOV technique. Eur J Radiol. 2011 Nov;80(2):e34-41. doi: 10.1016/j.ejrad.2010.06.038. Epub 2010 Jul 16. PMID 20638208
- [Background] Ma C, Li YJ, Pan CS, Wang H, Wang J, Chen SY, Lu JP. High resolution diffusion weighted magnetic resonance imaging of the pancreas using reduced field of view single-shot echo-planar imaging at 3 T. Magn Reson Imaging. 2014 Feb;32(2):125-31. doi: 10.1016/j.mri.2013.10.005. Epub 2013 Oct 18. PMID 24231348
- [Background] Riffel P, Michaely HJ, Morelli JN, Pfeuffer J, Attenberger UI, Schoenberg SO, Haneder S. Zoomed EPI-DWI of the pancreas using two-dimensional spatially-selective radiofrequency excitation pulses. PLoS One. 2014 Mar 3;9(3):e89468. doi: 10.1371/journal.pone.0089468. eCollection 2014. PMID 24594702
- [Background] Kim H, Lee JM, Yoon JH, Jang JY, Kim SW, Ryu JK, Kannengiesser S, Han JK, Choi BI. Reduced Field-of-View Diffusion-Weighted Magnetic Resonance Imaging of the Pancreas: Comparison with Conventional Single-Shot Echo-Planar Imaging. Korean J Radiol. 2015 Nov-Dec;16(6):1216-25. doi: 10.3348/kjr.2015.16.6.1216. Epub 2015 Oct 26. PMID 26576110